CLINICAL TRIAL: NCT01409902
Title: Using a Sheathed Speculum to Visualize and Access the Cervix In Women With Excessive Vaginal Tissue
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 105827
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Vaginal Prolapse
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main objective of the study is to assess the effectiveness of the sheathed speculum in providing adequate visualization and access to the cervix in patients with excessive vaginal tissue.

The secondary objective is to rate the patient's comfort evaluation during the sheathed speculum examination.

DETAILED DESCRIPTION:
This is a descriptive clinical trial designed to assess the efficacy of a sheathed speculum in providing adequate visualization and access to the cervix in women with excessive vaginal tissue. Eligible, consented subjects who fail their initial speculum examination (because their cervix is not visualized due to the collapse of loose lateral vaginal walls) will have a sheathed speculum examination instead of the standard-of-care exam whereby the clinician fabricates a solution at the bedside (condom with tip cut placed on speculum, concomitantly using an additional instrument like a lateral-wall retractor, glove with tip of thumb placed over the speculum, using the largest speculum available)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 64 years
* BMI greater than 30 (or see next line)
* Collapsing vaginal tissue preventing the visualization of the cervix (meeting this criterion in the absence of a BMI >30 would also qualify the patient for the study).
* Able to provide written informed consent

Exclusion Criteria:

* Patients unwilling to participate in the study or provide consent Presence of significant acute pelvic pain syndromes (ie exacerbation of dyspareunia, chronic pelvic pain or pelvic floor dysfunction, atrophic vaginitis, interstitial cystitis, endometriosis) which, in the opinion of the examining clinician, could potentially confound the patient's responses to the questionnaire
* Presence of active genital herpes
* Presence of significant condyloma acuminata (may be an investigator decision)
* Any other patient deemed inappropriate for the study by the consenting or examining investigator.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: excessive vaginal tissue
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2008-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adequate visualization and access to cervix or vaginal vault | At time of speculum exam

CONTACTS AND LOCATIONS:
Overall Officials: Erich Wyckoff, M, Principal Investigator — University of South Florida
Locations (1):
- USF STC, Tampa, Florida, United States